CLINICAL TRIAL: NCT00509314
Title: The Mechanism of Melanocyte Self-Assembly on Biomaterials and the Functional Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Other Study IDs: 9561703036
Record Dates: First submitted 2007-07-29; First posted 2007-07-31 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2006-05

CONDITIONS: Melanocyte; Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: melanocyte self-assembly and functional analysis

SUMMARY:
The aim of this study is to survey melanocytes in the ability of self-assembly on biomaterials and functional analysis in vitro. Also, this study may provide a better way for treatment of vitiligo after understanding the functional aspects of melanocytes.

DETAILED DESCRIPTION:
Vitiligo is a chronic disease that causes loss of melanocyte and pigment of the skin. Traditional treatments for vitiligo including topical corticosteroids and phototherapy lead to limited clinical effects. Autologous melanocyte transplantation is another way to treat vitiligo. However, the effect is largely affected by whether cultivated melanocytes are successfully uptaken by vitiliginous skin. The aim of this study is to survey the self-assembly on biomaterials and functional analysis. In the long run, this study may provide a better way for treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving cosmetic removal of moles

Exclusion Criteria:

* No special exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-05; Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Jan Lin, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Lin SJ, Jee SH, Hsaio WC, Lee SJ, Young TH. Formation of melanocyte spheroids on the chitosan-coated surface. Biomaterials. 2005 Apr;26(12):1413-22. doi: 10.1016/j.biomaterials.2004.05.002. PMID 15482829
- [Background] Lin SJ, Jee SH, Hsiao WC, Yu HS, Tsai TF, Chen JS, Hsu CJ, Young TH. Enhanced cell survival of melanocyte spheroids in serum starvation condition. Biomaterials. 2006 Mar;27(8):1462-9. doi: 10.1016/j.biomaterials.2005.08.031. Epub 2005 Sep 19. PMID 16171860